CLINICAL TRIAL: NCT01806844
Title: Cerebral Oxygenation During Resuscitation and Post-resuscitation Phase
Brief Title: Prehospital Cerebral Oxygenation During Cardiopulmonary Resuscitation (CPR)
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Cornelia Genbrugge, Dr. Genbrugge, Hasselt University
Other Study IDs: Copernicus I
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Cerebral oxygenation; Pre-hospital
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Near infrared spectroscopy (NIRS) is a technique that measures regional cerebral oxygenation in a non-invasive manner. Through the use of near infrared light, the difference between oxygenated and deoxygenated hemoglobin can be measured. By applying the Beer-Lamber law, a numeric result can be calculated. During a cardiac arrest, there is no stroke volume, no cardiac output and no cerebral perfusion. By using cerebral NIRS during out-of hospital cardiac arrest, low flow time and return of spontaneous circulation, this study wants to show the prognostic value of NIRS as extra monitoring.

ELIGIBILITY:
Inclusion Criteria:

* >16 year

Exclusion Criteria:

* DNR code

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pre-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
prognostic value | 1 year
  Prognostic value of cerebral oxygenation during CPR

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Genbrugge, MD, Principal Investigator — Hasselt University
Locations (5):
- Belgium (5):
  - Ziekenhuis netwerk Antwerpen, Antwerp, Antwerpen
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Universitair ziekenhuis Leuven, Leuven, Vlaams Brabant
  - GZA St Vincentius, Antwerp
  - AZ Turnhout, Turnhout

REFERENCES:
- [Background] Meex I, De Deyne C, Dens J, Scheyltjens S, Lathouwers K, Boer W, Vundelinckx G, Heylen R, Jans F. Feasibility of absolute cerebral tissue oxygen saturation during cardiopulmonary resuscitation. Crit Care. 2013 Mar 1;17(2):R36. doi: 10.1186/cc12546. PMID 23448653